CLINICAL TRIAL: NCT05990582
Title: Neurodevelopmental Outcomes and Morbidities of Moderate and Late Preterm Children at the Age of 9 Years -The Alkmaar MLPTI Cohort Study
Brief Title: The Alkmaar MLPTI Cohort Study: Outcomes at 9 Years
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Noordwest Ziekenhuisgroep (Other)
Responsible Party: Principal Investigator, F. (Femke) de Groof, Principal Investigator, MD, PhD, Noordwest Ziekenhuisgroep
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NL82197.029.22
Record Dates: First submitted 2023-07-25; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Preterm Birth; Developmental Delay; Growth Delay
Keywords: Moderate and late preterm infants; Neurodevelopmental outcomes; Growth; Morbidities
MeSH Terms: conditions — Premature Birth; Learning Disabilities; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: Outcomes of a group of preterm born children are compared to a group of children born at term.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MLPTI Cohort (Experimental): Group of 9 year old children born between 32 and 36 weeks of gestational age
  Interventions: Diagnostic Test: CBCL; Diagnostic Test: SDQ; Diagnostic Test: CCC-2-NL; Diagnostic Test: MCH Feeding scale; Diagnostic Test: TRF; Diagnostic Test: WISC-5-NL; Diagnostic Test: Movement ABC; Diagnostic Test: CELF-5-NL; Diagnostic Test: Emma Toolbox
- Control cohort (Active Comparator): Group of 9 year old children born at term
  Interventions: Diagnostic Test: CBCL; Diagnostic Test: SDQ; Diagnostic Test: CCC-2-NL; Diagnostic Test: MCH Feeding scale; Diagnostic Test: TRF; Diagnostic Test: WISC-5-NL; Diagnostic Test: Movement ABC; Diagnostic Test: CELF-5-NL; Diagnostic Test: Emma Toolbox

INTERVENTIONS:
Diagnostic Test: CBCL — A questionnaire on behaviour
  Other Names: Child Behaviour Checklist
Diagnostic Test: SDQ — A questionnaire on behaviour
  Other Names: Strength and Difficulties Questionnaire
Diagnostic Test: CCC-2-NL — A questionnaire on communcational skills
  Other Names: Children's Communication Checklist
Diagnostic Test: MCH Feeding scale — A questionnaire on feeding problems
  Other Names: Montreal Children's Hospital Feeding Scale
Diagnostic Test: TRF — A questionnaire on behaviour
  Other Names: Teacher report form
Diagnostic Test: WISC-5-NL — An IQ test for children
  Other Names: Wechsler Intelligence Scale of Development for Children
Diagnostic Test: Movement ABC — A test to assess motor function
  Other Names: MABC-II-NL
Diagnostic Test: CELF-5-NL — A test to assess language development
  Other Names: Clinical Evaluation of Language Fundamentals
Diagnostic Test: Emma Toolbox — Test of executive functions

SUMMARY:
Objective of the study:

To examine cognition, motor function, executive functions, speech and language development, behaviour, psychosocial functioning,academic achievement, physical morbidities and growth of MLPTI at the age of 9 years and correlate this with BSID-III-NL scores,growth parameters and body composition at the age of 2 years.

Study design:

This study will be a prospective open, non-therapeutic exploratory cohort study and can be seen as a continuation on the study with protocol identification number NL50800.094.14, performed in the NWZ Alkmaar between 2014 and 2016. This was a study on growth and neurodevelopment of MLPTI in the first 2 years of life.

Study population:

The study population is a group of 200 moderate and late preterm children who were born in the NWZ Alkmaar between 2014 and 2016. 100 of these children participated in the aforementioned study on growth and neurodevelopment at the age of 2 years. The oldest children in this group will reach the age of 9 years in 2023. Brothers/sisters/friends of these children aged between 8 and 10 will be asked as control group (n=50).

Primary study parameters/outcome of the study:

The main study parameters are the IQ-scores of the WISC-V, the motoric scores of the Movement-ABC, the executive functions of the EMMA Toolbox, the presence of morbidities, the growth pattern and the mean blood pressure at 9 years of age.

Secondary study parameters/outcome of the study:

Secondary outcome parameters are the he behavioural and psychosocial outcomes of the CBCL and the SDQ scores, speech-and language-developmental scores of the CELF-5-NL and CCC-2-NL, MCH Feeding Scale and Teacher Report Form (TRF) scores. Other outcome parameters are the relation between the 9-year outcomes and the BSID-III scores at the age of 2, and the differences between the MLPTI and the control group. Furthermore, we aim to determine the relation between growth and body composition in the first two years of life and the waist circumference, growth parameters and blood pressure at the age of 9 years.

DETAILED DESCRIPTION:
SUMMARY Rationale: Recent studies indicate that moderate and late preterm infants (MLPTI, gestational age (GA) 32-36 weeks) are at risk of lower IQ scores, behavioural and attention problems and academic underachievement at the age of 6 to 10 years. These recent findings of impaired outcomes above the age of 6 contrast with earlier studies that suggested that outcomes of MLPTI are comparable to those of full-term children. However, since the number of studies performed on MLPTI above 6 years of age is limited and show different results, the developmental outcomes of MLPTI remains a subject of debate and more research to this subject is warranted.

In addition, one recent study correlated impaired behavioural outcomes and lower IQ-scores at the age of 6 with the attentional and language scores of a Bayley Scales of Infant and Toddler Development (BSID-III) performed at the age of 1.5 to 2 years. This relation, however, is not confirmed in other studies. More research is therefore necessary to clarify the predictive value of these screening methods in early detection of impaired outcomes during school age, and to examine whether a longer follow-up could thereby help to prevent these problems.

Objective: To assess neurodevelopmental outcomes (including neurocognitive, motor, language, behavioral, and academic functioning), growth and morbidities in MLPTI children at the age of 9 born in the NWZ Alkmaar, and compare these outcomes to those of a sex and age-matched control group of friends of MLPTI children born at uncomplicated full term gestational age.

Study design: This study will be a prospective open, non-therapeutic exploratory cohort study and can be seen as a continuation on the study with protocol identification number NL50800.094.14, performed in the NWZ Alkmaar between 2014 and 2016. That study described growth, body composition and neurodevelopmental outcome of MLPTI in the first 2 years of life.

Study population: The study population is a group of 200 moderate and late preterm children who were born in the NWZ Alkmaar between 2014 and 2016. A total number of hundred children participated in the aforementioned study on growth and neurodevelopment at the age of 2 years. The oldest children of this cohort will reach the age of 9 years in January 2023. Sex and age-matched friends of these children whom are also 9 years old will be examined as control group of same aged peers (n=70).

Intervention: Parents will be asked to fill in five widely used questionnaires, including the Child Behaviour Checklist (CBCL), Strengths and Difficulties Questionnaire (SDQ), Childrens Communication Checklist (CCC-2-NL), Montreal Childrens Hospital Feeding Scale (MCH Feeding Scale) and a custom made questionnaire on morbidities. Teachers will be asked to complete the Teacher report form (TRF)), which is a version of the CBCL adapted for teachers. Children will visit the outpatient clinic once for neurodevelopmental assessment, including the Wechsler Intelligence Scale of Development for Children (WISC-V-NL) to assess intelligence (IQ), the EMMA-Toolbox to assess neurocognitive functioning, the Movement ABC (MABC-II-NL) to assess motor function, and subtests of the Clinical Evaluation of Language Fundamentals (CELF-5-NL) to assess language development. Furthermore, academic achievement will be assessed using existing data collected at school as part of the student monitoring system (National Institute for Educational Measurement (CITO)). During the same single visit, length, weight, waist circumference and blood pressure will be measured to analyse the body composition.

Main study parameters/endpoints: To examine neurodevelopmental outcomes (including neurocognitive, motor, language, and (eating-)behavioral function, and academic achievement), growth and morbidities in MLPTI children at the age of 9 born in the Noordwest Ziekenhuis, location Alkmaar, and compare them with a control group of 9 year old friends born at full term.

Secondary study parameters/outcome of the study:

Secondary outcome parameters are the he behavioural and psychosocial outcomes of the CBCL and the SDQ scores, speech-and language-developmental scores of the CELF-5-NL and CCC-2-NL, The Montreal Children Hospital feeding Scale and Teacher Report Form scores. Other outcome parameters are the relation between the 9-year outcomes and the BSID-III scores at the age of 2, and the differences between the MLPTI and the control group. Furthermore, we aim to determine the relation between growth and body composition in the first two years of life and the waist circumference, growth parameters and blood pressure at the age of 9 years.

.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all the following criteria:

* The participant is born in or transferred to the NWZ Alkmaar between January 1st, 2014 and April 18th, 2016 (the time in which the participants of trial NL50800.094.14 were born).
* The participant born at a gestational age from 32 to 35+6 weeks.
* Both parents of the participant have given informed consent to participate in the 9 years trial

In order to be eligible to participate in the control group of this study, a subject must meet all the following criteria:

* The participant is 9 years old when participating in this study and is a friend or classmate of the included MLPTI.
* Both parents of the participant have given informed consent for the participation of the study.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* The participant's parents are not able to fill out questionnaires or perform tests in Dutch.
* The participant has a severe developmental or genetic disorder and is thereby not able to perform the tests.
* The participant is not able to come to the outpatient clinic to do the tests.

A potential subject who meets any of the following criteria will be excluded from participation in this study as part of the control group:

* The participant is born with a GA < 37 weeks.
* The participant has a severe developmental or genetic disorder and is thereby not able to perform the tests.
* The participant had complications after birth (e.g. admission at a Neonatal ward)
* The participant needs special education

Ages: 9 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2023-08-06 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Full scale IQ | At 9 years of age
  The primary index scores and the FSIQ are on a standard score metric with a mean of 100 and an SD of 15. The primary index scores range from 45 to 155; the FSIQ ranges from 40 to 160.
  For both the primary index scores and the FSIQ, scores ranging from 90 to 109 are typically considered average
M-ABC score | At 9 years of age
  Standard Score: Total and percentile Total score 0, percentile 96-100 (high) Totalscore 4, percentile 54 (moderate) Totalscore 10, percentile 15 (consider help/intervention) totalscore 13,5, percentile 5 (intervention needed)
Executive functions on Emma-Toolbox | At 9 years of age
  Processing speed & Control Verbal Memory Visual memory Verbal working Memory Visual Working Memory Interpretation: Cortex. 2021 Oct;143:12-28. doi: 10.1016/j.cortex.2021.06.011. Epub 2021 Jul 14 Visuomotoric integration.
Prevalence of Morbidities | At 9 years of age
  This questionary scores the following morbities in percentages (numbers of participants with): re-admission in hospital, amount of infections, eczema, astma, speech and developmental problems, medication use, operations
Measurements of growth | At 9 years of age
  Length, weight, head and abdominal circumference are measured in cm. Parental height will be measured in cm.
Blood Pressure at 9 years of age | At 9 years of age
  Systolic bloodpressure in mmHg, range 5-200 Diastolic blood pressure in mmHg p-value is conducted for age.

SECONDARY OUTCOMES:
Behavioural and psychosocial outcomes of the CBCL | At 9 years of age
  Each item is scored using the scale: 0 = not true (as far as you know); 1 = somewhat or sometimes true; 2 = very true or often true. A total score of total behavorial problems is calculated and divided ingeTotal Score of behaviorial problems divided in internlizing behavorial problems and external behaviorial problems. A total T- score above 50 indicates that there are more problems than de controlgroup. the higher the score the more problems.
Speech- and language-developmental scores on CELF-5-NL | At 9 years of age
  Standard Score: This scores are derived from the total raw scores for each test and are on a normalized score scale that has a mean of 10 and a standard deviation (SD) of 3. A scaled score of 10 describes the average of a given age group. Scores of 7 and 13 are 1 SD below and above the mean, respectively The Children's Communication Checklist-2 U.S. Edition is a parent or caregiver rating scale based on the extensive research of author, Dr. Dorothy Bishop. CCC-2 helps rate aspects of communication, screens for general language, and identifies pragmatic language impairment. Domains that are tested is language: speech, syntax, sematics and coherence and pragmatics in scores.
  These scores are derived from the total raw scores for each test and are on a normalized score scale that has a mean of 10 and a standard deviation (SD) of 3 of 10 describes the average of a given age group. Scores of 7 and 13 are 1 SD below and above the mean, respectively
Children's Communication List CCC-2-NL | At 9 years of age
  The Children's Communication Checklist-2 U.S. Edition is a parent or caregiver rating scale based on the extensive research of author, Dr. Dorothy Bishop. CCC-2 helps rate aspects of communication, screens for general language, and identifies pragmatic language impairment. Domains that are tested is language: speech, syntax, sematics and coherence and pragmatics in scores.
  These scores are derived from the total raw scores for each test and are on a normalized score scale that has a mean of 10 and a standard deviation (SD) of 3 of 10 describes the average of a given age group. Scores of 7 and 13 are 1 SD below and above the mean, respectively
The Strengths and Difficulties Questionnaire (SDQ) | At age of 9 years
  The SDQ is a brief behavioural screening questionnaire about 2-17 year olds. It includes between one and three of the following components:
  A) 25 items on psychological attributes.
  All versions of the SDQ ask about 25 attributes, some positive and others negative. These 25 items are divided between 5 scales:
  1. emotional symptoms (5 items)
  2. conduct problems (5 items)
  3. hyperactivity/inattention (5 items)
  4. peer relationship problems (5 items)
  5. prosocial behaviour (5 items) A total score kan be calculated. A the T-score < 80 is considered as normal, 80-90 might indicate small problems,, a score > 90 indicates serious problems.
Teacher Report Form (TRH) | At 9 years of age
  This is the CBCL test filled in by the teacher. Each item is scored using the scale: 0 = not true (as far as you know); 1 = somewhat or sometimes true; 2 = very true or often true. A total score of total behavorial problems is calculated and divided ingeTotal Score of behaviorial problems divided in internlizing behavorial problems and external behaviorial problems. A total T- score above 50 indicates that there are more problems than de controlgroup. the higher the score the more problems.
Montreal Childrens Hospital Feeding Scale (MCH) | At 9 years of age
  The Montreal Children's Hospital Feeding Scale [MCH-Feeding Scale]) designed to identify feeding problems in children.
  Normal range = raw score 0-45 [T-score 35-60], mild difficulties = 46-52 [T-score 61-65], moderate 53-58 [T-score 66-70], severe >=59 [T-score >70].

CONTACTS AND LOCATIONS:
Overall Officials: METC AUMC, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Noordwest Ziekenhuisgroep, Alkmaar, Netherlands

IPD SHARING:
Plan to Share IPD: No